CLINICAL TRIAL: NCT00931346
Title: A Pilot Study of Pre-Exposure Prophylaxis (PrEP) to Evaluate Safety, Acceptability, and Adherence in At-risk Populations in Uganda, Africa
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: International AIDS Vaccine Initiative (Network)
Responsible Party: Patricia Fast MD PhD, Chief Medical Officer, International AIDS Vaccine Initiative
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IAVI E002
Record Dates: First submitted 2009-06-29; First posted 2009-07-02 (Estimated); Last update posted 2011-08-25 (Estimated); Status verified 2011-08

CONDITIONS: HIV Infection
Keywords: HIV; Human Immunodeficiency Virus
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- FTC/TDF Daily (Experimental): Daily dosing
  Interventions: Drug: FTC/TDF
- FTC/TDF Intermittent (Experimental): Dosed intermittently
  Interventions: Drug: FTC/TDF
- Placebo Daily (Placebo Comparator): Placebo dosed daily
  Interventions: Drug: Placebo
- Placebo Intermittent (Placebo Comparator): Placebo dosed intermittently, orally.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: FTC/TDF — emtricitabine/tenofovir disoproxil fumarate
  Arms: FTC/TDF Daily; FTC/TDF Intermittent
Drug: Placebo — Placebo
  Arms: Placebo Daily; Placebo Intermittent

SUMMARY:
This study will evaluate the safety and acceptability of intermittent and daily pre-exposure prophylaxis (PrEP) regimens with FTC/TDF (emtricitabine/tenofovir disoproxil fumarate) in HIV discordant couples, and it will directly compare adherence and intracellular drug levels in daily and intermittent PrEP recipients. It will also evaluate the relationship between drug adherence, sexual behavior and intracellular drug levels with an intermittent PrEP regimen. In addition it will evaluate the relationship between adherence to an intermittent PrEP regimen and timing of sexual activity in relation to PrEP dosing. The pilot will use objective medication event monitoring (MEMS) adherence measurement and evaluate the feasibility of newer adherence measurements such as hair sampling and plasma drug levels. This study will also evaluate the feasibility of using text messaging (SMS) to collect sexual activity data in an African setting. It will allow study teams and communities to prepare for potential subsequent larger trials of intermittent PrEP. The study is not sized to evaluate efficacy. If the intermittent PrEP regimen is safe, feasible in terms of adherence, and achieves intracellular drug levels similar to daily PrEP, the data could be used to design a larger phase 2 study with one or more intermittent PrEP regimens. The goal of such a larger trial would be to provide bridging data if daily PrEP regimens are found to be effective or to prepare for efficacy or non-inferiority trials of intermittent versus daily PrEP.

Investigation of immune responses associated with FTC/TDF will also be evaluated in the pilot study. The proportion of volunteers on FTC/TDF with HIV-specific immune responses, due to exposures that did not lead to established HIV infection, will be assessed at 2-3 time points and compared to responses in volunteers assigned to placebo. Immune responses may be correlated with risk behavior and host factors, such as human leukocyte antigen (HLA) type. As noted above, very few HIV infections are expected to occur during the study, so correlation of HIV-specific immune responses and protection from infection or attenuation of disease progression will not be possible until a larger study is conducted.

ELIGIBILITY:
Inclusion Criteria (for HIV-uninfected volunteers):

* Willing to comply with the protocol and available for follow-up for the study duration
* Has understood the information provided and has provided written informed consent before any study-related procedures are performed
* Willing to undergo couple HIV testing, sexually transmitted infection (STI) screening, HIV counseling and receive test results, and share results with partner
* At risk for HIV infection as defined by: has an HIV-infected partner not using ART in the past 3 months and had episodes of unprotected sex with partner in the past 3 months
* If a female of childbearing potential:

  * using an effective method of non-barrier contraception (hormonal contraceptive
  * intrauterine device (IUD)
  * surgical sterility) from 7 days prior to randomization until the end of the study
  * all female volunteers must be willing to undergo urine pregnancy tests
* HIV-infected partner is willing and eligible to enroll in the study

Inclusion Criteria (for HIV-1 infected partner):

* HIV-1 infected partner of an HIV-uninfected volunteer who meets study eligibility
* Plan to remain in the relationship for the duration of the study period
* Willing and able to provide written informed consent & locator information

Exclusion Criteria (for HIV-uninfected volunteer):

* Confirmed HIV-1 or HIV-2 infection
* Any clinically significant acute or chronic medical condition that is considered progressive, including severe infections requiring treatment such as tuberculosis, and alcohol or drug abuse
* Any of the following abnormal lab parameters:

  * Haemoglobin < 9.0 g/dL
  * Creatinine clearance <80mL/min, as calculated by Cockcroft-Gault equation
  * AST: > 2.5 x ULN
  * ALT: > 2.5 x ULN
  * Total bilirubin > 1.5 x ULN
  * Serum amylase > 1.5 x ULN
  * Serum phosphorus < 2.4 mg/dL
  * Urinalysis: Two abnormal dipsticks showing any of the following:

    * blood = 2+ or more (not due to menses);
    * protein = 1+ or more
    * leucocytes = 2+ or more
    * glucose= 1+ or more
* Confirmed diagnosis of chronic hepatitis B infection (HBsAg positive)
* If female, pregnant or planning a pregnancy within 4 months after enrolment or lactating
* Participation in another clinical study of a product currently, or within the 3 mo. prior to enrolment

Exclusion Criteria (for HIV-1 infected partner):

* Current use of antiretroviral therapy
* Concurrent enrollment in another HIV treatment trial

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2009-10; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability: volunteers with moderate and greater severity clinical adverse events, renal toxicities, and other moderate and severe laboratory abnormalities. | 6 months
Acceptability: proportion of volunteers who report willingness to use the study regimen; the acceptability to the HIV-infected partner of their partner using the investigational product | 6 months
Intracellular drug concentrations: the mean intracellular drug concentration for each group assigned to FTC/TDF | 6 months
Adherence: proportion of vol. who took, by MEMS data, at least 80% of doses; vol. assigned to FTC/TDF with detectable drug plasma levels within 48 hrs of use; relationship between intracellular drug levels and adherence in vol. assigned to FTC/TDF | 6 months
Behavioral: reported number of steady and casual sex partners; frequency of unprotected vaginal intercourse; substance use prior to or during sex | 6 months

SECONDARY OUTCOMES:
The proportion of volunteers who report somewhat high or high levels of burden in using electronic medication monitoring to measure adherence, and using cell phone communication to measure sexual activity | 6 months
The proportion of study days with missing SMS sexual activity data | 6 months
The proportion of volunteers assigned to placebo who have detectable intracellular drug levels | 6 months
The proportion of HIV-infected partners in discordant couples not on ART with detectable drug levels | 6 months
The proportion of volunteers with HIV-specific immune responses as measured by analysis of cellular or humoral immune response, or changes in gene regulation as measured by microarray or proteomic techniques | 6 months
The proportion of volunteers who report sharing medications | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Heiner Grosskurth, MD, Study Chair — MRC Entebbe; Anatoli Kamali, MD, Principal Investigator — MRC Entebbe
Locations (1):
- MRC-Entebbe, Entebbe, Entebbe, Uganda

REFERENCES:
- [Derived] Baxi SM, Liu A, Bacchetti P, Mutua G, Sanders EJ, Kibengo FM, Haberer JE, Rooney J, Hendrix CW, Anderson PL, Huang Y, Priddy F, Gandhi M. Comparing the novel method of assessing PrEP adherence/exposure using hair samples to other pharmacologic and traditional measures. J Acquir Immune Defic Syndr. 2015 Jan 1;68(1):13-20. doi: 10.1097/QAI.0000000000000386. PMID 25296098
- [Derived] Kibengo FM, Ruzagira E, Katende D, Bwanika AN, Bahemuka U, Haberer JE, Bangsberg DR, Barin B, Rooney JF, Mark D, Chetty P, Fast P, Kamali A, Priddy FH. Safety, adherence and acceptability of intermittent tenofovir/emtricitabine as HIV pre-exposure prophylaxis (PrEP) among HIV-uninfected Ugandan volunteers living in HIV-serodiscordant relationships: a randomized, clinical trial. PLoS One. 2013 Sep 26;8(9):e74314. doi: 10.1371/journal.pone.0074314. eCollection 2013. PMID 24086333
- See also: International AIDS Vaccine Initiative — http://www.iavi.org